CLINICAL TRIAL: NCT04610723
Title: Immunological Follow-up of Patients With Basedow's Orbitopathy : SIPO
Brief Title: Immunological Follow-up of Patients With Basedow's Orbitopathy
Acronym: SIPO
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL20_0597
Record Dates: First submitted 2020-10-26; First posted 2020-10-30 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2022-01

CONDITIONS: Graves Orbitopathy
Keywords: Graves orbitopathy; TRAK; Immune monitoring
MeSH Terms: conditions — Graves Ophthalmopathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — NC
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Graves' disease is characterized by the combination of anti-TSH receptor antibodies (Thyroid-Stimulating Hormone or thyroidotropic hormone), specific to this disease, with inconsistent symptoms such as hyperthyroidism, orbitopathy, goiter, or myxedema dermatological involvement. The activation of TSH receptors (RTSH) by these antibodies (known as "TRAK") causes the secretion of thyroid hormones as well as the development of the thyroid gland, responsible for a goiter. The cellular infiltrate responsible for the goiter consists mainly of T-lymphocytes but also of activated B lymphocytes secreting TRAK. Although Graves' disease is antibody mediated, cytokine secretion by Th1 therefore seems essential to pathogenesis. The treatment of orbitopathy requires primarily euthyroidism and the discontinuation of smoking. Despite these measures, moderate to severe attacks may require immunomodulatory treatment to limit local inflammation. This treatment is currently based on a first-line corticosteroid treatment (per os or preferably by weekly intravenous infusions). In the context of inadequate response, the therapeutic strategy is not very well established since some immunosuppressive treatments targeting B-cells or T- cells have been studied but with little benefit.

Many new concepts concerning immune tolerance and autoimmunity have emerged in recent years, particularly in Graves' disease, with sometimes complex cellular interactions. Certain mechanisms could occur either independently or in combination: i) modulation of T cell activation, differentiation and apoptosis; ii) inhibition of BL maturation and immunoglobulin production; iii) alteration of the balance between T helper (Th)-17 and T regulatory lymphocytes (Treg), by promoting Treg differentiation and inhibiting Th17 differentiation.

ELIGIBILITY:
Inclusion criteria:

* Patients aged 18 to 80 years included
* Subjects with Grave's disease and unsuccessful or intolerant to corticosteroid bolus therapy (EUGOGO protocol)
* Subjects with positive TRAKs

Exclusion criteria:

* Current treatment or within 6 months before inclusion by anti-CD20 monoclonal antibodies
* Current treatment or in the month prior to inclusion with corticosteroids >10 mg/day (oral or intravenous)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Graves' disease
Sampling Method: Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Quantify the subpopulations of CD4, CD8, Th, Treg and B-cells | 1 day
  Quantify the subpopulations of CD4, CD8, Th, Treg and B-cells in the peripheral blood of subjects with Graves' disease

SECONDARY OUTCOMES:
Compare the frequency and activation of lymphocyte subpopulations | 1 day
  Compare the frequency and activation of lymphocyte subpopulations in peripheral blood regarding TRAK levels
Compare the phenotypic characteristics of Tregs present | 1 day
  Compare the phenotypic characteristics of Tregs present in the peripheral blood of Graves' disease patients with Tregs in the peripheral blood of RA patients (previous laboratory data).

CONTACTS AND LOCATIONS:
Overall Officials: Yves-Marie PERS, MD,PhD, Study Director — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC